CLINICAL TRIAL: NCT02033408
Title: Manipulating the Microbiome in IBD by Antibiotics and Fecal Microbiota Transplantation (FMT): a Randomized Controlled Trial
Brief Title: Manipulating the Microbiome in IBD by Antibiotics and FMT
Acronym: FMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABCS-FMT-01
Record Dates: First submitted 2013-12-03; First posted 2014-01-10 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2019-04

CONDITIONS: Exacerbation of Ulcerative Colitis; Ulcerative Colitis, Active Severe; Crohn's Colitis
Keywords: IBD: Inflammatory Bowel Diseases; CD: Crohn's Disease; UC: Ulcerative Colitis; ASC: Acute Severe Colitis; FMT: Fecal Microbiota Transplantation; PUCAI: Pediatric Ulcerative Colitis Activity Index; Ciprofloxacin, Doxycycline, Gentamycin, amoxicillin, vancomycin, metronidazole,ciprofloxacin
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Anti-Bacterial Agents; Adrenal Cortex Hormones; Single Person

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antibiotics in addition to steroids (Experimental): methylprednisolone-1.5mg/kg up to 60mg daily in two divided doses and in addition the following antibiotics:
  1. PO Vancomycin 250mg 4 times a day for 3 weeks (children under age 8 125mgX4/d for 3 weeks)
  2. PO Amoxycillin 50mg per Kg divided by 3 (up to 500mg 3 times a day) - for 3 weeks
  3. PO Metronidazole 5mg per Kg 3 times a day (up to 250mg 3 times a day) - for 3 weeks
  4. PO Doxycycline 2mg per kg twice a day (up to 100mg twice a day) - for 3 weeks; OR- For children younger than 7 years: PO Ciprofloxacin 10mg per Kg twice a day (up to 250mg twice a day) for 3 weeks
  Interventions: Drug: AB (antibiotics)
- Steroids only (Active Comparator): methylprednisolone-1.5mg/kg up to 60mg daily in two divided doses
  Interventions: Drug: CS (corticosteroids) Only
- Open arm (Other): either the antibiotics and/or FMT (fecal microbiome transplant) may be administered in a non-randomized, uncontrolled open-label arm to any resistant IBD patients
  Interventions: Drug: AB (antibiotics); Drug: CS (corticosteroids) Only

INTERVENTIONS:
Drug: AB (antibiotics) — 1. PO Vancomycin 250mgX4/d for 3 weeks
  2. PO Amoxycillin 50mg/Kg divided by 3 (up to 500mgX3/d) - for 3 weeks
  3. PO Doxycycline 2mg/kg X2/d (up to 100mgX2/d) - for 3 weeks; OR- For children younger than 8 years: PO Ciprofloxacin 10mg/Kg X2/2 (up to 250mgX2/d) for 3 weeks
  Patients with known allergy to one of the drugs may be treated with oral Gentamycin (2.5mg/KgX3/d) for 3 weeks instead of the allergenic drug.
  Other Names: Ciprofloxacin-Ciprodex®; Doxycycline-Doxylin®; Gentamycin-Gentamicin®; Amoxicillin-Amoxyclav®; Vancomycin-Vanco-Teva®
  Arms: Antibiotics in addition to steroids; Open arm
Drug: CS (corticosteroids) Only — 1. methylprednisolone (1.5mg/kg up to 60mg daily in two divided doses)
  2. PO Metronidazole 5mg/Kg X3/d (up to 250mgX3/d) - for 3 weeks
  Other Names: Metronidazole-Flagyl®
  Arms: Open arm; Steroids only

SUMMARY:
the etiology of Inflammatory Bowel Diseases (IBD) is closely associated with the gut microbiome. The results of previous studies on the effectiveness of antibiotics and fecal macrobiota transplantation (FMT) are contradicting.

Aims: to evaluate the effectiveness of wide-spectrum antibiotic regimens in acute severe colitis in an addition to standard corticosteroid therapy (UC and isolated "UC-like" Crohn's colitis). The secondary aim is to assess the outcome of FMT in those not responding to five days of therapy (in either arm). As an exploratory aim, any IBD patient with a resistant disease to at least two immunosuppressive medications, may be treated with either interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children over the age the 2 years and adults of all ages with established diagnosis of UC using standard criteria (26, 27).
* Admission for IV steroid therapy
* PUCAI of at least 65 points at admission (i.e. severe attack)
* PUCAI>45 at enrollment
* Ability to swallow antibiotics (pills or syrup)

Exclusion Criteria:

* Change in dose or intervals of anti-TNF within the past 2 months prior to admission.
* Disease confined to the rectum (Proctitis).
* Antibiotic use in the past 4 weeks.
* Any known erosive inflammation anywhere in the small bowel or esophagus.
* Any proven infection such as positive stool culture, parasite or C. difficile, urinary tract infection, cellulitis, abscess, pneumonia, line-infections etc.
* Fever >38.5, or >38.0c thought to be unrelated to the inflammatory process of active UC.
* The probable need for second line medical therapy (infliximab, cyclosporine, tacrolimus) or colectomy within 5 days of enrollment, as judged by the caring physician.
* Known allergy to more than one antibiotic regimen from the list below.
* Pregnancy.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Total PUCAI (Pediatric Ulcerative Colitis Activity Index) score | at day 5 after treatment (compared between the two treatment groups).

SECONDARY OUTCOMES:
Remission rates | at days 7, separately at discharge, separately at day 14, and separately at 90 days.
  defined by PUCAI<10 without the need for second line therapy (anti TNF (Tumor Necrosis Factor), cyclosporine or tacrolimus) or colectomy.
Number of patients with PUCAI<35 points | at day 5
  without the need for second line therapy (anti TNF, cyclosporine or tacrolimus) or colectomy.
The need for second line therapy or colectomy by discharge | by 90 days and at 1 year
Rate of steroid | dependency at 1 year
  defined as a course longer than 3 month with an unsuccessful attempt to wean steroids or cumulative steroid treatment months of 4 months, during the year.
Need for subsequent admission | by 1 year
Calprotectin levels | at 5 and 14 days after treatment.
Rate of gastrointestinal carriage of resistant organisms (VRE, ESBL) | at days 5 and 14 after treatment.
Change in microbiome pattern. | 3 years from baseline
Rate of C. difficile infection | at days 5 and 14 after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Turner, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (12):
- The Hospital for Sick Children (SickKids), Toronto, Canada
- Hospital for Children and Adolescents Helsinki University Hospital, Helsinki, Finland
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Cener, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (2):
  - Università degli Studi di Napoli "Federico II", Napoli
  - Sapienza University of Rome, Rome
- Univeristy Children's Hospital in Krakow, Krakow, Poland
- Hospital Regional Universitario Carlos Haya Málaga, Málaga, Spain

REFERENCES:
- [Derived] Turner D, Bishai J, Reshef L, Abitbol G, Focht G, Marcus D, Ledder O, Lev-Tzion R, Orlanski-Meyer E, Yerushalmi B, Aloi M, Griffiths AM, Albenberg L, Kolho KL, Assa A, Cohen S, Gophna U, Vlamakis H, Lurz E, Levine A. Antibiotic Cocktail for Pediatric Acute Severe Colitis and the Microbiome: The PRASCO Randomized Controlled Trial. Inflamm Bowel Dis. 2020 Oct 23;26(11):1733-1742. doi: 10.1093/ibd/izz298. PMID 31833543